CLINICAL TRIAL: NCT06071689
Title: Radiographic Evaluation of the Peri-implant Circumferential Bone Level and Bone Changes in the Posterior Mandible of All-on-4 Implant Prosthesis With Different Materials and Bar Construction Techniques
Brief Title: Radiographic Evaluation of All-on-4 Implant Prosthesis With Different Materials and Bar Construction Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M0103023RP
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Bone Loss
Keywords: All-on-Four implant; PEEK framework; Soft metal; Selective laser melting
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEEK group (Active Comparator): patients receive all-on-4 prostheses constructed from CAD/CAM milled PEEK framework.
  Interventions: Device: screw retained prosthesis
- Soft metal group (Active Comparator): patients receive all-on-4 prostheses constructed from CAD/CAM milled soft metal framework.
  Interventions: Device: screw retained prosthesis
- selective laser melting group (Active Comparator): patients receive all-on-4 prostheses constructed from 3D printed selective laser melting Co-Cr framework.
  Interventions: Device: screw retained prosthesis

INTERVENTIONS:
Device: screw retained prosthesis — all-on-4 screw-retained prosthesis.
  Other Names: hybrid prosthsis

SUMMARY:
Eighteen patients will be selected from the outpatient clinic of the Prosthodontic Department, Faculty of Dentistry, Mansoura University seeking prosthetic rehabilitation.

patients will be randomly divided into three groups according to the framework materials: PEEK, Soft metal, and selective laser melting construction.

DETAILED DESCRIPTION:
All patients will receive conventional maxillary and mandibular complete dentures.

2. The mandibular denture will be modified by shortening the flanges and cutting the posterior part till the 1st molar then 3D scanned for recording the correct dimension of each tooth to be concerned during the construction of the superstructure and the final prosthesis.

3. Abutment level impression will be made, and the resultant cast will be 3D scanned for CAD/CAM construction of superstructure with abutments.

4. patients will be randomly divided into three groups according to the framework materials: PEEK, Soft metal, and selective laser melting construction.

5. The fit of the framework will be verified intraorally, and the final prosthesis will be digitally constructed; according to the dimensions of the scanned denture; to fit over the framework.

Evaluation Radiographic evaluation of circumferential bone level around implants and bone changes in the posterior mandible will be done using CBCT at one, two, three, and five years after insertion of the final prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous maxillary ridges and mandibular arch with four implants placed according to the All-on-4 distribution. All patients were recruited from the previous study.
* All selected patients will be with sufficient inter-arch space and restorative space.
* All selected patients will have healthy ridges covered by the compressible oral mucosa and free from any ridge flabbiness.

Exclusion Criteria:

* History of para-functional habits (Bruxism, clenching), smoking, and alcoholism.
* History of radiation therapy in the head and neck region.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
bone changes | 5 years
  circumferential peri-implant bone changes in mm

CONTACTS AND LOCATIONS:
Overall Officials: Khloud Ezzat, PhD, Principal Investigator — Lecturer
Locations (1):
- Khloud Ezzat, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mourad KE, Rashed NHAH, Altonbary GY, Fattah Hegazy SA. Five years of radiographic evaluation for the peri-implant bone changes of all-on-four implant prostheses constructed from different framework materials using different digital construction techniques. BMC Oral Health. 2024 Aug 7;24(1):910. doi: 10.1186/s12903-024-04642-7. PMID 39112988